CLINICAL TRIAL: NCT04969419
Title: Incidence of Melanoma and Non-melanoma Skin Cancer in People With Vitiligo: A Case-control Study in the United Kingdom, 2009-2020
Brief Title: Incidence of Melanoma and Non-melanoma Skin Cancer in People With Vitiligo
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: P045
Record Dates: First submitted 2021-07-01; First posted 2021-07-20 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Vitiligo; Melanoma (Skin); Nonmelanoma Skin Cancer; Squamous Cell Carcinoma; Basal Cell Carcinoma; Actinic Keratoses
MeSH Terms: conditions — Vitiligo; Melanoma; Carcinoma, Squamous Cell; Carcinoma, Basal Cell; Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a confirmed diagnosis of Vitiligo within the study period will be included as cases for analysis.
  Interventions: Other: Exposure of skin cancer of interest
- Controls: The controls will be defined by matching cases with people who have never been diagnosed with vitiligo either prior to or during the study period, by age and sex, at General Practice level.
  Interventions: Other: Exposure of skin cancer of interest

INTERVENTIONS:
Other: Exposure of skin cancer of interest — Melanoma and nonmelanoma skin cancers: squamous cell carcinoma, basal cell carcinoma and actinic keratoses.

SUMMARY:
This study examines melanoma and nonmelanoma skin cancer in people diagnosed with vitiligo compared to matched controls.

DETAILED DESCRIPTION:
For the primary analysis, this study examines the risk of melanoma and nonmelanoma skin cancers: squamous cell carcinoma and basal cell carcinoma in people diagnosed with vitiligo. It also examines actinic keratoses. In secondary analysis, this study examines the prevalence of skin cancer in people diagnosed with vitiligo compared to matched controls.

This study also examines whether the susceptibility to melanoma and nonmelanoma skin cancer may vary between different patient subgroups, e.g. ethnicity, those who undergo phototherapy or treatment with the new targeted biologic immunosuppressive therapies.

ELIGIBILITY:
Inclusion Criteria:

* All eligible adult patients (aged ≥ 18) registered with General Practioner (GP) practices contributing data to OPCRD between January 1, 2010 and December 31, 2020, were eligible for inclusion in the study. People diagnosed with vitiligo prior to the study period (prevalent vitiligo) and people newly diagnosed with vitiligo during the study period (incident vitiligo) are included as cases.

Exclusion Criteria:

* People actively registered with the GP practice at that date without a history of vitiligo require a minimum one-year registration with their GP practice.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will use routinely collected and collated data from Optimum Patient Care Research Database (OPCRD) to provide a broadly representative sample of the population of the UK.
Sampling Method: Non-Probability Sample
Enrollment: 75771 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data Ltd
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
OPCRD data can be accessed by bone fide researchers for specific research projects, subject to approval by Anonymised Data Ethics & Protocol Transparency (ADEPT) Committee. The data utilised for this study cannot be made available without such approval.
Supporting Information: Study Protocol
Time Frame: The data will be available subject to approvals for two years after the study publication date
Access Criteria: Data sharing is subject to ADEPT committee approval

REFERENCES:
- [Result] Ferguson J, Eleftheriadou V, Nesnas J. Risk of Melanoma and Nonmelanoma Skin Cancer in People with Vitiligo: United Kingdom Population-Based Cohort Study. J Invest Dermatol. 2023 Nov;143(11):2204-2210. doi: 10.1016/j.jid.2023.04.013. Epub 2023 May 3. PMID 37146674
- See also: Main publication of final results — https://doi.org/10.1016/j.jid.2023.04.013

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Controls
Started | 15156 | 60615
Completed | 15156 | 60615
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 15156 | 60615 | 75771
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [35 to 61] | 47 [35 to 61] | 47 [35 to 61]
Age, Customized [Count of Participants; unit: Participants]
  18-44 | 6724 | 26843 | 33567
  45-64 | 5393 | 21596 | 26989
  65+ | 3,039 | 12,176 | 15215
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8,256 | 33,016 | 41272
  Male | 6,900 | 27,599 | 34499
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8,049 | 32,196 | 40245
  Asian or Asian British | 2,067 | 6,096 | 8163
  Black or Black British | 345 | 1,272 | 1617
  Mixed | 155 | 557 | 712
  Not stated | 367 | 1,685 | 2052
  Other | 618 | 2,725 | 3343
  Missing data | 3555 | 16084 | 19639
Index of Multiple Deprivation [Median (Inter-Quartile Range); unit: Quintile of deprivation] — Index of Multiple Deprivation (IMD) is a UK national deprivation measure of deprivation which is based on the patient postcode. IMD has been stratified into quintiles with IMD 1 representing most deprived and IMD 5 being the least deprived.
  Quintile of deprivation | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of New Onset Skin Cancer in Adult People Diagnosed With Vitiligo
Description: Number of new onset skin cancer assessed prospectively in vitiligo cases and matched controls. The skin cancer outcome comprises of the composite of melanoma and nonmelanoma skin cancers: squamous cell carcinoma and basal cell carcinoma.
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 14982 | 59057
Participants | 133 | 812

2. Primary Outcome: Number of New Onset Skin Cancers in the Female Sex Subgroup
Description: Number of new onset skin cancers assessed prospectively in female vitiligo cases and matched controls.
Time Frame: 10 years from the index date
Population: The number of participants analyzed for this outcome is a subset of the overall population: female sex subgroup
Measure: Count of Participants; unit: Participants
Groups:
- Female Cases: Female patients with a confirmed diagnosis of Vitiligo within the study period will be included as cases for analysis.
  Exposure of skin cancer of interest: Melanoma and nonmelanoma skin cancers: squamous cell carcinoma, basal cell carcinoma and actinic keratoses.
- Female Controls: The controls will be defined by matching cases with people who have never been diagnosed with vitiligo either prior to or during the study period, by age and sex, at General Practice level.
  Exposure of skin cancer of interest: Melanoma and nonmelanoma skin cancers: squamous cell carcinoma, basal cell carcinoma and actinic keratoses.
Arm/Group | Female Cases | Female Controls
Number analyzed (Participants) | 8159 | 32121
Participants | 78 | 429

3. Primary Outcome: Number of New Onset Skin Cancers in the Male Sex Subgroup
Description: Number of new onset skin cancers assessed prospectively in male vitiligo cases and matched controls.
Time Frame: 10 years from the index date
Population: The number of participants analyzed for this outcome is a subset of the overall population: male sex subgroup
Measure: Count of Participants; unit: Participants
Groups:
- Male Cases: Male patients with a confirmed diagnosis of Vitiligo within the study period will be included as cases for analysis.
  Exposure of skin cancer of interest: Melanoma and nonmelanoma skin cancers: squamous cell carcinoma, basal cell carcinoma and actinic keratoses.
- Male Controls: The controls will be defined by matching cases with people who have never been diagnosed with vitiligo either prior to or during the study period, by age and sex, at General Practice level.
  Exposure of skin cancer of interest: Melanoma and nonmelanoma skin cancers: squamous cell carcinoma, basal cell carcinoma and actinic keratoses.
Arm/Group | Male Cases | Male Controls
Number analyzed (Participants) | 6823 | 26936
Participants | 55 | 383

4. Primary Outcome: Number of New Onset Skin Cancers in the <45 Age Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those aged <45
Time Frame: 10 years from the index date
Population: The number of participants analyzed for this outcome is a subset of the overall population:age less than 45 years subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6711 | 26789
Participants | 11 | 72

5. Primary Outcome: Number of New Onset Skin Cancers in the 45-64 Age Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those aged 45-64
Time Frame: 10 years from the index date
Population: The number of participants analyzed for this outcome is a subset of the overall population:age 45 tp 64 years subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 5,342 | 21,079
Participants | 42 | 315

6. Primary Outcome: Number of New Onset Skin Cancers in the >=65 Age Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those aged >=65
Time Frame: 10 years from the index date
Population: The number of participants analyzed for this outcome is a subset of the overall population:age 65+ years subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 2,929 | 11,189
Participants | 80 | 425

7. Primary Outcome: Number of New Onset Skin Cancers in the White Ethnicity Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those of white ethnicity
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 7932 | 31118
Participants | 103 | 563

8. Primary Outcome: Number of New Onset Skin Cancers in the Non-white Ethnicity Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those of non-white ethnicity
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 3179 | 12663
Participants | 9 | 66

9. Primary Outcome: Number of New Onset Skin Cancers in the Most Deprived Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those in the most deprived subgroup category
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 7681 | 30325
Participants | 46 | 345

10. Primary Outcome: Number of New Onset Skin Cancers in the Least Deprived Subgroup
Description: Number of new onset skin cancers assessed prospectively in vitiligo cases and matched controls by those in the least deprived subgroup category
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 5918 | 23307
Participants | 66 | 355

11. Secondary Outcome: Prevalence of Skin Cancer in Adult People Diagnosed With Vitiligo
Description: Skin cancer is defined as the composite of melanoma and nonmelanoma skin cancers: squamous cell carcinoma and basal cell carcinoma.
Time Frame: At index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6360 | 25439
Participants | 66 | 293

12. Secondary Outcome: Prevalence of Melanoma Skin Cancer in Adult People Diagnosed With Vitiligo
Description: Prevalence of melanoma skin cancer in adult people diagnosed with vitiligo at or before recruitment
Time Frame: At index date.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6360 | 25439
Participants | 85 | 27

13. Secondary Outcome: Prevalence of Squamous Cell Carcinoma Skin Cancer in Adult People Diagnosed With Vitiligo
Description: Prevalence of squamous cell carcinoma skin cancer in adult people diagnosed with vitiligo at or before recruitment
Time Frame: At index date.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6360 | 25439
Participants | 13 | 72

14. Secondary Outcome: Prevalence of Basal Cell Carcinoma Skin Cancer in Adult People Diagnosed With Vitiligo
Description: Prevalence of basal cell carcinoma skin cancer in adult people diagnosed with vitiligo at or before recruitment
Time Frame: At index date.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6360 | 25439
Participants | 31 | 161

15. Secondary Outcome: Number of New Onset Actinic Keratoses in Adult People Diagnosed With Vitiligo
Description: Number of new onset actinic keratoses in adult people assessed in vitiligo cases and matched controls.
Time Frame: 10 years from the index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 14896 | 58618
Participants | 264 | 1108

16. Secondary Outcome: Prevalence of Actinic Keratoses in Adult People Diagnosed With Vitiligo
Description: Prevalence of actinic keratoses in adult people diagnosed with vitiligo at or before recruitment
Time Frame: At index date.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 6360 | 25439
Participants | 111 | 363

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for the study.
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04969419/Prot_SAP_000.pdf